CLINICAL TRIAL: NCT02001207
Title: Association of Salivary Cortisol Levels and Outcome of Critically Ill Patients in the Intensive Care Unit
Brief Title: Salivary Cortisol in Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-1304-072-482
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2013-12

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MICU patients
  Interventions: Other: Salivary cortisol test

INTERVENTIONS:
Other: Salivary cortisol test

SUMMARY:
In critical illness, patients are highly stressed and should have elevated cortisol (stress hormone) secretion to adapt to stress. Dysfunction of this system is referred to as critical illness-related corticosteroid insufficiency. Free cortisol (unbound form) which is mainly responsible for its physiologic function is difficult to measure. We hypothesized that the salivary cortisol, which can be obtained by noninvasive methods, can more accurately evaluate adrenal function of critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who agreed to participate

Exclusion Criteria:

* Known adrenal or pituitary disease
* oral bleeding
* currently on systemic or inhaled corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit in Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | 28 days

SECONDARY OUTCOMES:
ICU days | 28 days
ventilator-free days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Min Lee, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea